CLINICAL TRIAL: NCT04994106
Title: A Phase I Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD5462 Following Single and Multiple Ascending Dose Administration to Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD5462 Following Single and Multiple Ascending Dose Administration to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: D9090C00001
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants
Keywords: Healthy participants of Japanese descent; First-in-Human; 2-part study

STUDY DESIGN:
Intervention Model Description: This is randomized single-blind, and placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is single blind with regard to treatment (AZD5462 or placebo). This means that the Principal Investigator, all clinical staff involved in the clinical study (except for the unblinded Pharmacist), the participants, and the site monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Cohort A1: AZD5462 Dose 1 (Experimental): Randomized healthy participants will receive Dose 1 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort A2: AZD5462 Dose 2 (Experimental): Randomized healthy participants will receive Dose 2 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort A3: AZD5462 Dose 3 (Experimental): Randomized healthy participants will receive Dose 3 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort A4 Japanese descent: AZD5462 Dose 3 (Experimental): Randomized participants of Japanese descent will receive Dose 3 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort A5: AZD5462 Dose 4 (Experimental): Randomized healthy participants will receive Dose 4 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort A6 Japanese descent: AZD5462 Dose 4 (Experimental): Randomized participants of Japanese descent will receive Dose 4 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort A7: AZD5462 Dose 5 (Experimental): Randomized healthy participants will receive Dose 5 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort A8 Japanese descent: AZD5462 Dose 5 (Experimental): Randomized participants of Japanese descent will receive Dose 5 of AZD5462.
  Interventions: Drug: AZD5462
- Part A: Placebo (Healthy Participants) (Placebo Comparator): Randomized healthy participants will receive Placebo matched to AZD5462.
  Interventions: Drug: Placebo
- Part A: Placebo (Japanese descent participants) (Placebo Comparator): Randomized participants of Japanese descent will receive Placebo matched to AZD5462.
  Interventions: Drug: Placebo
- Cohort B1: AZD5462 Dose 1 (Experimental): Randomized healthy participants will receive Dose 1 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort B2: AZD5462 Dose 2 (Experimental): Randomized healthy participants will receive Dose 2 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort B3: AZD5462 Dose 3 (Experimental): Randomized healthy participants will receive Dose 3 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort B4: AZD5462 Dose 4 (Experimental): Randomized healthy participants will receive Dose 4 of AZD5462.
  Interventions: Drug: AZD5462
- Cohort B5 Japanese descent: AZD5462 Dose 4 (Experimental): Randomized participants of Japanese descent will receive Dose 4 of AZD5462.
  Interventions: Drug: AZD5462
- Part B: Placebo (Healthy participants) (Placebo Comparator): Randomized healthy participants will receive Placebo matched to AZD5462.
  Interventions: Drug: Placebo
- Part B: Placebo (Japanese descent participants) (Placebo Comparator): Randomized participants of Japanese descent will receive Placebo matched to AZD5462.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5462 — Participants will receive AZD5462, at dose levels of 1 to 5 in part A and at 1 to 4 in part B, respectively.
  Arms: Cohort A1: AZD5462 Dose 1; Cohort A2: AZD5462 Dose 2; Cohort A3: AZD5462 Dose 3; Cohort A4 Japanese descent: AZD5462 Dose 3; Cohort A5: AZD5462 Dose 4; Cohort A6 Japanese descent: AZD5462 Dose 4; Cohort A7: AZD5462 Dose 5; Cohort A8 Japanese descent: AZD5462 Dose 5; Cohort B1: AZD5462 Dose 1; Cohort B2: AZD5462 Dose 2; Cohort B3: AZD5462 Dose 3; Cohort B4: AZD5462 Dose 4; Cohort B5 Japanese descent: AZD5462 Dose 4
Drug: Placebo — Participants will receive Placebo matched to AZD5462.
  Arms: Part A: Placebo (Healthy Participants); Part A: Placebo (Japanese descent participants); Part B: Placebo (Healthy participants); Part B: Placebo (Japanese descent participants)

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetic (PK) of AZD5462 following single ascending dose (SAD) and multiple ascending dose (MAD) administration in healthy male and female participants and healthy participants of Japanese descent.

DETAILED DESCRIPTION:
This Phase I, First in Human (FIH), randomized single-blind, placebo-controlled study will consist of 2 parts (Part A and Part B) with an interleaved study design.

Part A of the study will be a sequential SAD design with 5 dose levels planned to be investigated across 8 cohorts, of which 3 cohorts will solely comprise of participants of Japanese descent. Within each cohort, 6 participants will be randomized to receive AZD5462 and 2 participants randomized to receive placebo.

Part B of the study will be a sequential MAD design with 4 dose levels of AZD5462 planned to be investigated across 5 cohorts, of which 1 cohort will comprise solely of participants of Japanese descent. Within each cohort 6 participants will be randomized to receive AZD5462 and 2 participants randomized to receive placebo.

The duration for participants randomized to Part A of the study is 5 to 6 weeks, and for Part B, 6 to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) participants aged 18 to 50 years of age and healthy participants of Japanese descent, 20 to 50 years of age, with suitable veins for cannulation or repeated venipuncture
* Females must have a negative pregnancy test at the Screening Visit
* Have a body mass index between 18 and 32 kg/m^2 inclusive and weigh at least 50 kg and no more than 105 kg inclusive
* For cohorts comprised solely of participants of Japanese descent, a participant will be considered of Japanese descent only if both parents and all grandparents are Japanese

Exclusion Criteria:

* History of any clinically important disease or disorder
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study drug
* Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results
* Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody, and Human immunodeficiency virus
* Abnormal vital signs
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5462
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of study drug
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days (or 5 half-lives, whichever is the longest) of the first administration of study drug in this study
* Clinical signs and symptoms consistent with Coronavirus disease 2019, eg, fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening or on admission

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Upto Follow-up (Part A: Day 10 ± 3; Part B: Day 19 ± 3)
  Assessment of the safety and tolerability of AZD5462 following administration of single ascending doses (Part A) and multiple ascending doses (Part B).

SECONDARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) for AZD5462 | Part A: Day 1 (pre-dose and post-dose), and Days 2, 3, and 10 (post-dose); Part B: Days 1 to 19 (pre and post-doses)
  Characterization of the single dose and steady state PK of AZD5462 following administration.
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) for AZD5462 | Part A: Day 1 (pre-dose and post-dose), and Days 2, 3, and 10 (post-dose); Part B: Days 1 to 19 (pre and post-doses)
  Characterization of the single dose and steady state PK of AZD5462 following administration.
Area under plasma concentration time curve from zero to infinity (AUCinf) for AZD5462 | Part A: Day 1 (pre-dose and post-dose), and Days 2, 3, and 10 (post-dose); Part B: Days 1 to 19 (pre and post-doses)
  Characterization of the single dose and steady state PK of AZD5462 following administration.
Renal clearance of drug from plasma (CLR) for AZD5462 | Part A: Day 1 (pre-dose and post-dose), and Days 2, 3, and 10 (post-dose); Part B: Days 1 to 19 (pre and post-doses)
  Characterization of the single dose and steady state PK of AZD5462 following administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home